CLINICAL TRIAL: NCT04184544
Title: Supporting Women and Girls in Pakistan: Scaling up Empowerment and Care Strategies to Address Health and Survival
Brief Title: Scaling up Evidence Based MNCH Interventions : A Quasi Experimental Study Umeed e Nau (UeN) Project
Acronym: UeN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor and Founding Director, Aga Khan University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 0979-3131
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Maternal Complication of Pregnancy; Newborn Morbidity; Perinatal Problems

STUDY DESIGN:
Intervention Model Description: Implementation research to Scale up of evidence based interventions comprising four components 1) Designing of management protocol and revision of training curricula and Capacity building of outreach and facility based health care providers; 2) sustained supplies of essential drugs and commodities; 3) community engagement through Lady health worker program and 4) Health Management information data improvement and use of the data for decision making to improve provision and quality of services
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal and Newborn health districts (Experimental): Group one included maternal and newborn health districts. These districts are further divided into three sub groups. Sub group 1 will receive only interventions focusing on maternal health (1 district (Sangher)); sub group 2 will receive interventions focusing only on newborn health (1 district (Nasirabad)); sub group 3 will receive combined maternal and newborn interventions (two districts (, Lasbila and Badin).
  Interventions: Other: Improving of quality of care at health facility and outreach level
- Child Health (Experimental): Group two will receive child health interventions focusing on the implementation of the global action plan for pneumonia and diarrhea (GAPPD [4districts, Qamabar Shahdadkot Muzaffargarh, Rahim Yar Khan Jafferabad).
  Interventions: Other: Improving of quality of care at health facility and outreach level

INTERVENTIONS:
Other: Improving of quality of care at health facility and outreach level — Community Mobilization and engagement; Use of DHIS data for decision making; Capacity building of health care workers and providers and other Community level and facility level interventions to improve MNCH outcomes

SUMMARY:
The Umeed-e-Nau (UeN) initiative aims to support the introduction, scale up, and further piloting of high quality and high impact interventions to improve Maternal, Newborn And Child Health (MNCH)in Pakistan by harnessing the potential of both public and private sectors, coupled with introduction of women and girls empowerment interventions. UeN has two major components: 1) Introducing proven effective MNCH interventions at scale in 8 rural districts of Pakistan, and 2) Generating evidence on innovative approaches to improve MNCH while included in public health programs in Pakistan. There are six trials that are being conducted to address different evidences gaps to improve maternal, newborn and child health in Pakistan. The protocols of the trials will be registered separately.

DETAILED DESCRIPTION:
Pakistan's continued high maternal, neonatal, and child mortality is affecting the overall development and national growth. The estimated national maternal mortality ratio ranges from 250 - 750 per 100,000 live births per year, while neonatal mortality rate ranges from 43 - 66 per 1,000 live births per year across the provinces of Pakistan. The under-five mortality rate is 89 per 1,000 live births per year, and diarrhea and pneumonia are two of the most common causes of post-neonatal mortality. Together, they account for more than 30% of all under five deaths in Pakistan.

Majority of maternal, newborn and child deaths are preventable and treatable given programs are designed and delivered through an efficient public health system that takes into account the geographic and social structures. There are several factors resulting in slow progress and improvement of MNCH indicators. These include poor coverage, delayed scale up of effective interventions within the existing health system platforms, lack of women's and girls' empowerment, voice, and participation, and lack of community awareness and support regarding health conditions and poverty. Many of the risk factors that impact maternal and newborn health, such as nutritional deficiencies, exist from adolescence, and becoming pregnant during this sensitive life stage has been found to slow and stunt one's growth In order to evaluate the impact of the UeN initiative quasi experimental study design will be used. The intervention groups are broadly divided into two groups. Both groups will serve as control against each other due to nature of targeting of age group by each intervention group type. Group one included maternal and newborn health districts. These districts are further divided into three sub groups. Sub group 1 will receive only interventions focusing on maternal health (1 district (Sangher)); sub group 2 will receive interventions focusing only on newborn health (1 district (Nasirabad)); sub group 3 will receive combined maternal and newborn interventions (two districts (Lasbila and Badin). Group two will receive child health interventions focusing on the implementation of the global action plan for pneumonia and diarrhea (GAPPD [4districts, Qamabar Shahdadkot Muzaffargarh, Rahim Yar Khan Jafferabad). This design will help us to evaluate independent and combined effect of maternal, newborn, and child health interventions to address maternal, newborn and child health outcomes. We hypothesize that the roll out of proven and effective interventions within existing health delivery platforms for maternal, newborn, child and adolescent health will lead to significant reduction in perinatal mortality rate (20% compared to baseline) and at least 30% reduction in diarrhea and pneumonia case fatality rate in the target project districts.

UeN design justification: The conceptual framework for UeN postulates that increased engagement with communities, empowering women and girls, including addressing access barriers; 2) strengthening capacity of the public and private health sectors mainly through revision of curricula based on new evidence, developing management protocols for different cadre of health workers and providers on MNCH and training; private Sector engagement; 3) provision of sustained supplies and 4) District Health Information System (DHIS) data use for decision making will lead to greater responsiveness of public and private service providers to women's and girls' needs - particularly those of undeserved women, girls and children. The UeN initiative aims to create opportunities in governance processes through revival and participation in District Health Management team (DHMTs), service delivery and citizens' voice and empowerment to transform public and private health sector interactions to drive improvements in MNCH and survival

ELIGIBILITY:
Inclusion Criteria:

* All women of reproductive age in the project areas
* All children under the age of five years

Exclusion Criteria:

* The subjects not residing in the project catchment population

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal deaths | three years
  20% reduction in perinatal mortality
case fatality rate | Three years
  30% reduction in Pneumonia and diarrhea case fatality in participating health facilities

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, PhD, Principal Investigator — AKU
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muhammad S, Memon ZA, Mian A, Wasan Y, Rizvi A, Ahmed I, Soofi S, Cousens S, Bhutta ZA. A cross-sectional analysis of the impact of lady health worker visits in the prenatal and postnatal period on the uptake of continuum of care interventions and childhood mortality in Pakistan. J Glob Health. 2025 Jun 2;15:04158. doi: 10.7189/jogh.15.04158. PMID 40452336
- [Derived] Memon ZA, Muhammad S, Soofi S, Khan N, Akseer N, Habib A, Bhutta Z. Effect and feasibility of district level scale up of maternal, newborn and child health interventions in Pakistan: a quasi-experimental study. BMJ Open. 2020 Jul 14;10(7):e036293. doi: 10.1136/bmjopen-2019-036293. PMID 32665387